CLINICAL TRIAL: NCT05909761
Title: An Observational Pregnancy Safety Study in Women With Neuromyelitis Optica Spectrum Disorder (NMOSD) Exposed to UPLIZNA® (Inebilizumab-cdon) During Pregnancy
Brief Title: Observational Safety Study in Women With Neuromyelitis Optica Spectrum Disorder (NMOSD) Exposed to UPLIZNA® During Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: VIB0551.P4.S4; EUPAS105613 (Other: European Union Post Authorization Studies)
Expanded Access: NCT06590051 (Available)
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorder; Pregnancy Related
Keywords: Neuromyelitis Optica Spectrum Disorder; Pregnancy; UPLIZNA; inebilizumab; birth complications
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: UPLIZNA — Enrolled female participants with NMOSD who were exposed to UPLIZNA during pregnancy will be assessed. No study drug will be administered.
  Other Names: inebilizumab-cdon

SUMMARY:
This is an observational study to monitor female participants exposed to UPLIZNA during pregnancy. This study requires voluntary reporting of pregnancies in female participants with NMOSD exposed to UPLIZNA during pregnancy or within 6 months preceding conception. Pregnancy-related data, potential confounding factors and information related to pregnancy outcome will be collected. The schedule of office visits and all treatment regimens will be determined by the treating healthcare provider. Duration of the study is 10 years, at minimum.

DETAILED DESCRIPTION:
Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Are a female of reproductive potential with a confirmed or suspected diagnosis of NMOSD
* Have been exposed to UPLIZNA during pregnancy as defined by receipt of any dose during pregnancy or within 6 months preceding conception

Note: Other Protocol Defined Inclusion/Exclusion Criteria Apply

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will consist of participants who have been exposed to UPLIZNA during pregnancy and have signed an informed consent form (ICF).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2032-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of newborns with Major Congenital Malformations (MCMs) | Minimum of 10 years
Number of newborns with Preterm birth | Minimum of 10 years
Number of newborns with low birth weight | Minimum of 10 years
Number of stillbirths | Minimum of 10 years

SECONDARY OUTCOMES:
Number of newborns with Minor Congenital Malformations | Minimum of 10 years
Number of infants with developmental milestone abnormalities | Minimum of 10 years
Number of infants with neurologic abnormalities | Minimum of 10 years
Number of infants with immune system development abnormalities | Minimum of 10 years
Number of Spontaneous Abortions | Minimum of 10 years
Number of Induced or Elective Abortions | Minimum of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com